CLINICAL TRIAL: NCT02457676
Title: Improving Self Regulation in Children With Fetal Alcohol Syndrome Spectrum Disorders: A Neuroplastic Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Joanne Rovet, Senior Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000014076
Record Dates: First submitted 2014-11-19; First posted 2015-05-29 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Fetal Alcohol Spectrum Disorders
Keywords: Self-Regulation Training; Neuroimaging; Response Inhibition; Behavioral Regulation; Emotional Regulation
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alert Program for Self-Regulation (Experimental): Participants with FASD who received the Alert Program for Self-Regulation therapy between the two testing periods.
  Interventions: Behavioral: Alert Program for Self-Regulation
- FASD Alert Waitlist (No Intervention): Participants with FASD who did not receive therapy between the two testing periods but were provided intervention on study completion.
- Typically Developing Control (No Intervention): Normally developing controls not exposed to alcohol in utero who were not treated between the two testing periods.

INTERVENTIONS:
Behavioral: Alert Program for Self-Regulation — Children attend 12 1.5 hour weekly sessions. Alert uses the analogy of a car engine to help children identify their own self-regulatory behavior. Children learn strategies to regulate their own "engine speed" in different situations.
  Arms: Alert Program for Self-Regulation

SUMMARY:
This study on children with fetal alcohol spectrum disorder (FASD) aims to (i) characterize their self-regulation deficits, a process important for controlling emotions and behavior, (ii) describe brain structure and function underlying self-regulation, and (iii) determine whether training to improve self-regulation abilities changes brain and behavior. Individuals with FASD have a high risk of cognitive and social deficits, which reflect their difficulties in self-regulation and may lead to mental health concerns in adulthood. Importantly, early intervention improves long-term outcome. However the full extent of self-regulation problems in FASDs is unknown and the underlying neuroanatomy has not been fully described. Furthermore, information on how to best treat children with FASDs is lacking. Thus, the investigators propose three studies with a sample of 8-12 year old children, 40 with FASDs and 20 typically developing controls. In Study 1, the participants will be evaluated on cognitive and social self-regulation abilities using clinical and experimental tests. In Study 2, the participants will undergo a 1-hour MRI scanning session to obtain measures of their brain structure and function. In Study 3, FASDs will be randomly assigned to an immediate or delayed treatment group. The immediate group will undergo 12-weeks of therapy with the Alert Program for Self Regulation®. On conclusion of training, all will repeat Studies 1 and 2 and following this retest, the delayed treatment group will undergo training. The investigators will evaluate change in cognitive and social behavior and in brain structure and function by comparing performance and neuroimaging findings before and after the intervention. The investigators expect Alert training to significantly improve behavior and alter brain regions important for self-regulation. The findings will yield important information for improving self-regulation in FASDs and mitigating the development of mental health challenges.

ELIGIBILITY:
Inclusion Criteria:

* FASD: diagnosis of FAS/pFAS or ARND OR
* healthy child

Exclusion Criteria:

* head injury or other neurological abnormality
* debilitating or chronic medical condition affecting the nervous system
* MRI contraindication, such as braces
* inability to read
* non-English speaking
* IQ below 80 (typically developing controls only)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2009-10; Primary Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Emotion regulation | 14 weeks after initial testing
  Evaluated by parent questionnaires

SECONDARY OUTCOMES:
Inhibitory control: Test of Everyday Attention for Children; NEPSY, BRIEF | 14 weeks after initial testing
  Evaluated by neuropsychological tests
Social cognition: Saltzman's Social Cognitive Task; NEPSY | 14 weeks after initial testing
  Evaluated by neuropsychological tests
Behavior: Behavior Rating Inventory of Executive Function; Child Behavior Checklist | 14 weeks after initial testing
  Evaluated by parent questionnaires
Brain structure: Voxel-based morphometry | 14 weeks after initial testing
  Voxel-based morphometry analyses
Brain structure: Cortical thickness | 14 weeks after initial testing
  Civet pipeline
Brain function: Functional MRI | 14 weeks after initial testing
  Response inhibition paradigm

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Rovet, PhD, Principal Investigator — The Hospital for Sick Children

REFERENCES:
- [Result] Soh DW, Skocic J, Nash K, Stevens S, Turner GR, Rovet J. Self-regulation therapy increases frontal gray matter in children with fetal alcohol spectrum disorder: evaluation by voxel-based morphometry. Front Hum Neurosci. 2015 Mar 4;9:108. doi: 10.3389/fnhum.2015.00108. eCollection 2015. PMID 25788884
- [Result] Nash K, Stevens S, Greenbaum R, Weiner J, Koren G, Rovet J. Improving executive functioning in children with fetal alcohol spectrum disorders. Child Neuropsychol. 2015;21(2):191-209. doi: 10.1080/09297049.2014.889110. Epub 2014 Jul 10. PMID 25010354